Validation of the Screening Instrument: PRISMA-7 for Frailty among Elderly Hospitalized Danes

Date: 20.06.2019

ID REG-070-2017

# **Background**

The demographic development with an increasing proportion of elderly persons makes it necessary to develop instrument that may be used to identify those individuals who are in need of a more intensive support from the health and social systems in order to prevent morbidity, loss of function or hospitalization. The British Geriatric Society recommend using PRISMA-7 for screening among elderly community dwelling adults in order to identify frail elderly persons in need of a more comprehensive geriatric assessment (1). PRISMA-7 was developed in Canada as part of a project aiming to identify and improve treatment of elderly persons with loss of function. The acronym stands for Program of Research to Integrate the Services for the Maintenance of Autonomy (2-3). PRISMA-7 has been validated I Germany (4) and in Holland (5) but to our knowledge not in Denmark.

## Aim

The aim of this study is to validate a Danish version of PRISMA-7.

#### Methods

PRISMA-7 was translated in to Danish and back translated into English and disagreements hereafter resolved. Patients 75 years or older who were dismissed from a hospital stay and by the hospital physiotherapist were considered to need further physical training in the municipality after dismissal were screened with PRISMA-7. This was done successively in the period May 1<sup>st</sup> 2017 until December 31<sup>st</sup> 2018. Data on individual PRISMA scores were stored in an EasyTrial Database.

## Statistical methods

Every Danish Citizen has a unique personal identification number. This makes it possible to follow every person included in our study and assess mortality, morbidity, use of health services in the community, and use of medications (6-8). In regression models, we will study possible associations between PRISMA-7 scores and mortality, morbidity, and use of health services.

## **Ethics**

In Denmark registry studies are not requested to be approved by the ethical committee. This study was approved by the Danish Data Protection authorities. The EasyTrial database used for storage of PRISMA-7 results is approved by Region Zealand as a safe place to store individual data. Any use of the EasyTrial database is logged.

- 1. Turner, G. and A. Clegg, Best practice guidelines for the management of frailty: a British Geriatrics Society, Age UK and Royal College of General Practitioners report. Age Ageing, 2014. **43**(6): p. 744-7.
- 2. Hebert, R., et al., *Frail elderly patients. New model for integrated service delivery.* Can Fam Physician, 2003. **49**: p. 992-7.
- 3. Raiche, M., R. Hebert, and M.F. Dubois, *PRISMA-7: a case-finding tool to identify older adults with moderate to severe disabilities.* Arch Gerontol Geriatr, 2008. **47**(1): p. 9-18.
- 4. Braun, T., C. Gruneberg, and C. Thiel, *German translation, cross-cultural adaptation and diagnostic test accuracy of three frailty screening tools : PRISMA-7, FRAIL scale and Groningen Frailty Indicator.* Z Gerontol Geriatr, 2018. **51**(3): p. 282-292.
- 5. Hoogendijk, E.O., et al., *The identification of frail older adults in primary care: comparing the accuracy of five simple instruments.* Age Ageing, 2013. **42**(2): p. 262-5.

- 6. Lynge, E., J.L. Sandegaard, and M. Rebolj, The Danish National Patient Register. Scand J Public Health, 2011. **39**(7 Suppl): p. 30-3.
- Andersen, J.S., F. Olivarius Nde, and A. Krasnik, *The Danish National Health Service Register*. 7. Scand J Public Health, 2011. **39**(7 Suppl): p. 34-7. Kildemoes, H.W., H.T. Sorensen, and J. Hallas, *The Danish National Prescription Registry*. Scand J
- 8. Public Health, 2011. **39**(7 Suppl): p. 38-41.